CLINICAL TRIAL: NCT01461902
Title: Measuring Vasospasm, Biomarkers, and Neurocognitive Outcomes in Pediatric Traumatic Brain Injury
Brief Title: Vasospasm in Pediatric Traumatic Brain Injury
Acronym: PTBI
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00027860
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Brain Injury
Keywords: traumatic brain injury; brain injury; head injury; vasospasm
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pediatric Traumatic Brain Injury: Children from 5 days to 15 years of age who have been admitted to the hospital with a traumatic brain injury.

SUMMARY:
The purpose of this study is to assess for vasospasm using Transcranial Doppler (TCD) and brain injury biomarkers, and evaluate neurocognitive outcome data in pediatric traumatic brain injury (TBI) patients who have experienced a mild to severe head injury.

ELIGIBILITY:
Inclusion Criteria:

1. admission to Duke University Children's Hospital;
2. age 5 days to 15 years;
3. a diagnosis of a TBI with a GCS 3-15;
4. capable of adequate TCD ultrasound examination;
5. and presence of intravenous or arterial access (blood) and/or an EVD for cerebrospinal fluid (CSF) and/or Foley catheter/ability to void unassisted (urine) biomarker collection unless they are excluded based on the exclusion criteria.

Exclusion Criteria:

* the presence of previously diagnosed significant neurodevelopmental delay,
* a diagnosis of non-traumatic intracranial hemorrhage and
* parents/legal guardians who do not speak or understand English.

Ages: 5 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients who have been admitted for a traumatic brain injury to Duke University Hospital.
Sampling Method: Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-09; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Vasospasm detection by Transcranial Doppler Ultrasound | 8 days
  Daily transcranial doppler ultrasound performed in pediatric traumatic head injury patients.

SECONDARY OUTCOMES:
Detection of biomarkers in pediatric traumatic brain injury | 2 days
  Detection of a defined set of protein biomarkers from biological samples collected upon enrollment, 12, 24, and 48 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Reuter-Rice, PhD, Principal Investigator — Duke University School of Nursing and School of Medicine
Locations (1):
- Duke University medical Center, Durham, North Carolina, United States